CLINICAL TRIAL: NCT04300881
Title: Treatment of Post-Ocriplasmin Therapy Vitreolysis Induced Subretinal Fluid With Eplerenone (Mineralocorticoid Antagonists): The TOTEM Study
Brief Title: Treatment of Post-Ocriplasmin Therapy Vitreolysis Induced Subretinal Fluid With Eplerenone (Mineralocorticoid Antagonists)
Acronym: TOTEM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment
Sponsor: Wagner Macula & Retina Center (Other)
Collaborators: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WM562718
Record Dates: First submitted 2019-11-21; First posted 2020-03-09 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Vitreomacular Traction; Subretinal Edema
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Eplerenone
  Interventions: Drug: Eplerenone
- Control (No Intervention)

INTERVENTIONS:
Drug: Eplerenone — Following intravitreal ocriplasmin therapy
  Arms: Treatment

SUMMARY:
Evaluate the efficacy of eplerenone as an adjunctive treatment to intravitreal ocriplasmin for subretinal fluid in comparison to a control group of only receiving intravitreal ocriplasmin in patients with symptomatic vitreomacular adhesion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Symptomatic VMA, VMT, or macular hole
* BCVA 20/30 - CF 3' Snellen equivalent
* Willing and able to provide signed informed consent and willing to undertake all scheduled study-related assessments, visits, and treatments
* JETREA® treatment naïve

Exclusion Criteria:

* Patients who are pregnant, planning to become pregnant, or breastfeeding a child
* Uncontrolled ocular hypertension or glaucoma in study (defined as IOP ≥ 25mm Hg or a cup to disc ratio (CDR) > 0.8 despite treatment with anti-glaucoma medication)
* Active malignancies within the last 12 months except appropriately treated carcinoma in situ of the crevices, melanoma, and prostate cancers treated with a curative intent
* Inability to comply with study or follow-up procedures
* Women who may become pregnant or lactating or intend to become pregnant during the study
* Known drug allergy to ocriplasmin or eplerenone
* Patients with known contraindications Eplerenone as outlined in the package insert

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Central Foveal Thickness (CFT) over time | through study completion, an average of 1 year
  Changes as assessed via SD-OCT from the lowest CST measurement in the study, due to disease activity

SECONDARY OUTCOMES:
Changes from baseline in Best Corrected Visual Acuity (BCVA) over time | through study completion, an average of 1 year
  Changes as assessed using the visual acuity chart at a starting distance of 4 meters

CONTACTS AND LOCATIONS:
Locations (1):
- Wagner Macula & Retina Center, Norfolk, Virginia, United States